CLINICAL TRIAL: NCT06432569
Title: Evaluation of Butyrate and Palmitoylethanolamide Effects on Intestinal Permeability and Microbiota Gut Composition in Patients With Irritable Bowel Syndrome - A Double-blind, Placebo-controlled Crossover Randomized Study
Brief Title: Evaluation of Butyrate and Palmitoylethanolamide in IBS Patients (B/P3_1)
Acronym: B/P3_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5475-AO-22
Record Dates: First submitted 2023-02-27; First posted 2024-05-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome With Diarrhea

STUDY DESIGN:
Intervention Model Description: The study has two arms: Group 1: n=25 Treatment A e Group 2: n=25 Treatment B (with - Treatment A: 3 capsules/day of butyrate (625 mg) + 3 capsules/day PEA (200 mg) at a ratio of dosage of 3/1 - Treatment B: Placebo (3+3/day capsules of starch).
  Eligible subjects with IBS will be randomized in a 1:1 ratio to the treatment A or treatment B for six weeks. After the first treatment period, there is a 14-day washout period.
  Hence, individuals will be treated with B/A treatment for additional six weeks, according to the crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ButirBioma+PeaBioma (Active Comparator): Treatment : 3 capsules/day of butyrate (625 mg) + 3 capsules/day PEA (200 mg) at a ratio of dosage of 3/1
  Interventions: Dietary Supplement: ButirBioma + PeaBioma
- Placebo (Placebo Comparator): Treatment Placebo :(3+3/day capsules of starch).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ButirBioma + PeaBioma — randomized in a 1:1 ratio to treatment Butir+Pea or treatment with Placebo for six weeks. After the first treatment period, there is a 14-day washout period.
  Arms: ButirBioma+PeaBioma
Dietary Supplement: Placebo — Placebo( 3+3 cps/die)
  Arms: Placebo

SUMMARY:
Evaluation of the effects of butyrate ( BitirBioma) and palmitoylethanolamide( PEA=PeaBioma) on intestinal permeability and gut microbiota composition in patients with irritable bowel syndrome.

Study B/P 3_1 is an interventional study involving the use of food supplements on the market (BitirBioma Plus and PeaBioma Plus), single-center, double-blind, placebo-controlled, crossover, randomized, in n=50 patients with bowel syndrome irritable, diarrheal and mixed variant (IBS-D and IBS-M), lasting for one year.

The study has two arms: Group 1: n=25 Treatment A e Group 2: n=25 Treatment B (with - Treatment A: 3 capsules/day of butyrate (625 mg) + 3 capsules/day PEA (200 mg) at a ratio of dosage of 3/1 - Treatment B: Placebo (3+3/day capsules of starch).

Eligible subjects with IBS will be randomized in a 1:1 ratio to treatment A or treatment B for six weeks. After the first treatment period, there is a 14-day washout period.

Hence, individuals will be treated with B/A treatment for additional six weeks, according to the crossover design.

In the two treatment periods, subjects will be required to complete a visual analogue score VAS questionnaire to assess gastrointestinal symptoms and Stool Bristol Scales. During the visit, the subjects will have to record Questionnaire Rome IV to evaluate their quality of life. At the same time, it will be theirs required to provide:

* fecal sample for the evaluation of the composition of fecal microbiota (Biomaplan Kit)
* a urine sample for the evaluation of intestinal permeability (Gastropack) a capillary blood sample and a serum sample for the detection of Zonulin (Kit Healthy gut and Immundiagnostik AG )
* a capillary blood sample and a serum sample for the detection of Zonulin (Kit Healthy gut and Immundiagnostik AG )

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory condition affecting the colon, characterized by relapsing and remitting mucosal inflammation. It presents with symptoms like bloody diarrhea, rectal urgency, fatigue, and abdominal pain. While various therapies are available for managing UC, including medications like amino salicylates, corticosteroids, immunomodulators, and biologics, there's ongoing research into supportive treatments like probiotics.

Probiotics are beneficial microorganisms that can positively influence gut health by modifying the gut microbiota, improving intestinal barrier function, and balancing immune response. Several studies have investigated their efficacy in UC management. Notably, the probiotic mixture VSL#3, containing strains of Lactobacillus and Bifidobacteria, has shown promising results in inducing remission in UC patients.

Other probiotic products like E. coli Nissle 1917, L. rhamnosus GG, and L. casei DG have also demonstrated effectiveness in maintaining disease remission or prolonging relapse-free periods in UC patients. The product Prolife 10 FORTE, containing multiple strains of Lactobacillus, Bifidobacteria, and Bacillus coagulans, along with prebiotic components and vitamins, has shown potential in positively influencing gut microbiota composition and metabolic activity in healthy individuals.

Based on these promising findings, further investigation is warranted to evaluate the potential of Prolife 10 FORTE in improving the gut microbiota composition of UC patients during the remission phase.

ELIGIBILITY:
Inclusion Criteria:

* ● IBS patients (both males and females) with positive diagnosis based on Rome IV criteria (IBS-D and IBS-M)

  * Age in the range 18-70 years
  * Subjects capable of conforming to the study protocol
  * Subjects who have given their free and informed consent

Exclusion Criteria:

-Any relevant organic, systemic or metabolic disease, including celiac disease, IDDM (Insulin- Dependant Diabetes Mellitus), Insulin-Independent Diabetes Mellitus, metabolic syndrome, pelvic organ prolapses, urinary incontinence, ulcerative colitis, Crohn's disease, microscopic colitis, infectious colitis, ischemic colitis, complicated diverticular disease.

* Subjects with untreated food intolerance, i.e. remaining symptomatic despite the withdrawal of the suspected food
* Prior major gastrointestinal surgeries
* Females of childbearing potential, in the absence of effective contraceptive methods
* Subjects who become unable to conform to protocol
* Subjects who are continuously taking contact laxatives
* Subjects who are treated continuously with glucocorticoids, anti-histaminergic and mast cell stabilizer drugs
* Subjects who are treated continuously with trimebutine
* Recent history or suspicion of alcohol abuse or drug addiction
* Subjects who are treated with antibiotics or probiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the variation of gut microbiota composition (Microbiota test ) | 9 months
  Collection of faecal sample for the assessment of the faecal microbiota composition ( rRNA16S) The 16S rRNA gene is a bacterial ribosomal gene and a part of the 30S subunit which is used in the identification, characterization, and classification of various bacteria. Samples were normalized, pooled, and run on Illumina MiSeq , in order to evaluate the composition of gut microbiota in terms of bacterial diversity ( alfa and beta) and abundance and any variability associated with the treatment.

SECONDARY OUTCOMES:
Evaluation of intestinal permeability(4 sugar test: Gastropack) | 12 months
  1. Analysis of mannitol( normal range 15-25%), lactulose( n.r. 0,45%-0,75%), sucrose(normal < 0,15%) and sucralose( normal<1,5%); L/M (normal <0.03%; borderline 0,03%-0,09%; >0.09 severe):
  2. a capillary blood sample for the detection of Zonulin (Healthy gut Kit) )/Immundiagnostik AG )( normal cut-off 6-10 ng/mL)
Evaluation of Gastrointestinal symptoms( questionary) | 4 months
  Every evening during the two treatment periods, subjects must record a VAS(Visual Analogue Scale : 1-10; 1= non pain; 10= worst pain possible) questionnaire to assess gastrointestinal symptoms and the Stool Bristol Scale.( 1-7; normal 3-4)
Evaluation of Quality of Life (IBS-SSS score) (questionary) | 4 months
  At the visit time points, subjects will have to record the IBS-SSS score( points 75-174 mild, 175-300 moderate; >300 severe)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Savarino, Prof,MD, Principal Investigator — University of Padova
Locations (1):
- Edoardo Vinvenzo Savarino, Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: No